CLINICAL TRIAL: NCT00511407
Title: A Multi-Center, Randomized, Phase II Study To Assess Safety and Efficacy With the Renal Assist Device (RAD) In Patients With Acute Renal Failure
Brief Title: Open-Label Study To Evaluate the Safety and Efficacy of the Renal Assist Device In Patients With Acute Renal Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RenaMed Biologics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD-002
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Acute Renal Failure
Keywords: Acute renal failure; Bioartificial kidney; Cell therapy; Hemofiltration; Septic shock
MeSH Terms: conditions — Acute Kidney Injury; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): RAD Treatment
  Interventions: Device: Renal tubule assist device
- II (No Intervention): Conventional CVVHD

INTERVENTIONS:
Device: Renal tubule assist device — Standard hemofiltration cartridge containing nonautologous human renal tubule cells, connected to conventional continuous venovenous hemodialysis circuit.
  Arms: I

SUMMARY:
Although conventional hemodialysis removes waste products and corrects fluid imbalance, it does not replace critical absorptive, metabolic, endocrine, and immunologic functions performed by healthy renal tubule cells. This trial involving patients with acute renal failure evaluates the efficacy and safety of an extracorporeal renal assist device (RAD) containing human renal tubule cells connected to a conventional hemodialysis circuit. It is hypothesized that short-term (72-h) use of this cell therapeutic device will improve survival of ARF patients compared to patients receiving only conventional continuous renal replacement therapy.

DETAILED DESCRIPTION:
Acute Renal Failure (ARF) is a severe inflammatory disease state often accompanied by Multi-Organ Failure (MOF) and Systemic Inflammatory Response Syndrome (SIRS). ARF is precipitated by many factors and is most often linked to the loss of kidney tubule cell function. Patients with ARF are treated in the intensive care units of hospitals, and recovery of renal function is vitally important to their survival. Current therapy for ARF involves conventional kidney support with continuous renal replacement therapies (CRRT). Despite advances in treating patients with CRRT, ARF has an extremely high mortality rate (55-70%) and requires extensive hospital stays, predominantly in the ICU. The RAD is designed to both treat ARF with MOF and/or SIRs and facilitate the natural recovery of a patient's own kidney function. The RAD is intended for use for short periods of time in conventional extracorporeal therapeutic systems that are already available in the hospital. The RAD therapy operates outside the body and is designed to mimic the structure and function of the natural kidney. In this manner it is intended to replace the missing metabolic, endocrine, and immunologic functions of the kidney and allow time for the patient's own kidneys to resume normal functions.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant.
* Requiring continuous renal replacement therapy for treatment of acute renal failure secondary to acute tubular necrosis in ICU setting.
* At least one non-renal organ failure or presence of sepsis.

Exclusion Criteria:

* Contraindications to systemic anticoagulation with heparin.
* Irreversible brain damage.
* Presence of any organ transplant.
* Presence of preexisting chronic renal failure prior to this episode of acute renal failure.
* Acute renal failure occurring in the setting of burns, obstructive uropathy, allergic interstitial nephritis, acute or rapidly progressive glomerulonephritis, vasculitis, hemolytic-uremic syndrome, thrombotic thrombocytopenic purpura (TTP), malignant hypertension, scleroderma renal crisis, atheroembolism, functional or surgical nephrectomy, hepatorenal syndrome, cyclosporine or tacrolimus nephrotoxicity.
* Metastatic malignancy which is actively being treated or may be treated by chemotherapy or radiation during the subsequent three month period after RAD therapy.
* Chronic immunosuppression.
* Receiving Xigris therapy at time of randomization.
* Severe liver failure as documented by a Pugh Liver Failure Score.
* Do Not Resuscitate (DNR) status.
* Platelet count 35,000/mm3 within 4 hours of platelet transfusion.
* Patient not expected to survive 28-days because of an irreversible medical condition.
* Any medical condition that the investigator thinks may interfere with the study objectives.
* Concurrent enrollment in another clinical trial that could affect the outcome of this study protocol.
* Use of any other Investigational drug or device within the previous 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 28, 90, and 180 d
Time to recovery of renal function | 180 d
Time to ICU and hospital discharge | 180 d

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of Alabama, Birmingham, Alabama
  - Medical College of Georgia, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Western New England Renal and Transplant Associates, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Southeast Renal Associates/Presbyterian Hospital, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia